CLINICAL TRIAL: NCT02854410
Title: Dietary Nitrate on Salivary Flow for Nasopharyngeal Carcinoma Patients Pre and Post Concurrent Chemo-radiation Therapy
Brief Title: Dietary Nitrate on Salivary Flow for Nasopharyngeal Carcinoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Songlin Wang, Professor and Vice President of Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: changsm2005
Record Dates: First submitted 2016-07-23; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: dietary sodium nitrate; radiotherapy; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — sodium nitrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium nitrate supplementation (Experimental): Patients will receive Sodium nitrate supplementation from 7 days before radiotherapy to one month after the end of radiotherapy
  Interventions: Dietary Supplement: Sodium nitrate
- Placebo Comparator(sodium chloride) (Placebo Comparator): Patients will receive placebo from 7 days before radiotherapy to one month after the end of radiotherapy
  Interventions: Dietary Supplement: sodium chloride

INTERVENTIONS:
Dietary Supplement: Sodium nitrate — Dietary intake:Sodium nitrate 0.5mmol/kgbodyweight,bid
  Arms: Sodium nitrate supplementation
Dietary Supplement: sodium chloride — Dietary intake:sodium chloride 0.5mmol/kgbodyweight,bid
  Arms: Placebo Comparator(sodium chloride)

SUMMARY:
The purpose of this study is to evaluate whether dietary nitrate supplementation could improve the salivary flow for nasopharyngeal carcinoma patients receiving concurrent chemo-radiation therapy.

DETAILED DESCRIPTION:
Thirty patients diagnosed as nasopharyngeal carcinoma will be recruited. Nitrate supplement(Sodium nitrate: 0.5 mmol/kgbodyweight,bid) or placebo(sodium chloride: 0.5 mmol/kgbodyweight,bid) will be provided to the patients from 7 days before radiotherapy to one month after the finish of radiotherapy . The salivary flow and plasma nitrate levels will be determined before the course of nitrate supplementation and radiotherapy,before the course of radiotherapy,post the course of radiotherapy immediately and one month after the finish of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed stages III-IVb (UICC 2002) nasopharyngeal carcinomas, will be recruited.

Exclusion Criteria:

* Patients with local invasion or metastatic foci in salivary glands, detected by MRI and positron emission computed tomography(PET-CT) prior to treatment, were excluded, as were patients suffering from diseases, such as Sjogren's syndrome, or with a history of surgery to major salivary glands, or prior head and neck radiotherapy.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change of salivary flow | one day before the course of nitrate supplementation and radiotherapy,one day before the course of radiotherapy,one day post the course of radiotherapy and one month after the finish of radiotherapy

SECONDARY OUTCOMES:
Chang of plasm nitrate level | one day before the course of nitrate supplementation and radiotherapy,one day before the course of radiotherapy,one day post the course of radiotherapy and one month after the finish of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Wang Songlin, PHD, Study Chair — Capital Medical University shool of stomatology
Locations (1):
- Capital Medical University School of Stomatology, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xia DS, Deng DJ, Wang SL. Destruction of parotid glands affects nitrate and nitrite metabolism. J Dent Res. 2003 Feb;82(2):101-5. doi: 10.1177/154405910308200205. PMID 12562881
- [Background] Xia DS, Liu Y, Zhang CM, Yang SH, Wang SL. Antimicrobial effect of acidified nitrate and nitrite on six common oral pathogens in vitro. Chin Med J (Engl). 2006 Nov 20;119(22):1904-9. PMID 17134590
- [Background] Xia D, Deng D, Wang S. Alterations of nitrate and nitrite content in saliva, serum, and urine in patients with salivary dysfunction. J Oral Pathol Med. 2003 Feb;32(2):95-9. doi: 10.1034/j.1600-0714.2003.00109.x. PMID 12542832
- [Background] Bryan NS, Ivy JL. Inorganic nitrite and nitrate: evidence to support consideration as dietary nutrients. Nutr Res. 2015 Aug;35(8):643-54. doi: 10.1016/j.nutres.2015.06.001. Epub 2015 Jun 11. PMID 26189149
- [Background] Xia D, Qu X, Tran SD, Schmidt LL, Qin L, Zhang C, Cui X, Deng D, Wang S. Histological characteristics following a long-term nitrate-rich diet in miniature pigs with parotid atrophy. Int J Clin Exp Pathol. 2015 Jun 1;8(6):6225-34. eCollection 2015. PMID 26261499